CLINICAL TRIAL: NCT06453005
Title: Comparative Evaluation of SMART Hall Technique Versus Conventional SS Crown Restoration in Treatment of Carious Primary Molars - a Randomized Clinical Trial
Brief Title: Comparative Evaluation of SMART Hall Technique Vs. Conventional SS Crown in Primary Molars: a Randomized Clinical Trial
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C K S Teja Institute Of Dental Sciences & Research (Other)
Responsible Party: Principal Investigator, P K Saraswathi Bai, Post Graduate Student, C K S Teja Institute Of Dental Sciences & Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKSTeja
Record Dates: First submitted 2024-05-25; First posted 2024-06-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Caries,Dental; Pain; Plaque, Dental; Gingival Bleeding
Keywords: Randomized Clinical Trial; Dental caries; Primary molars; Stainless Steel Crowns; SMART Hall Technique; Conventional Technique; Silver Diamine Fluoride; Split Mouth Study
MeSH Terms: conditions — Dental Caries; Pain; Dental Plaque; Gingival Hemorrhage

STUDY DESIGN:
Intervention Model Description: Our study involves comparing two different dental treatment modalities (SMART Hall technique and standard SSC restoration) in a split-mouth design, where each participant serves as their control, the Single group model aligns with the structure of your study. This model indicates that all participants receive the intervention(s) being studied, which is consistent with our split-mouth study design.
Masking Description: Participants are masked to treatment allocation, while care providers and investigators are not. Outcomes assessors remain masked to minimize bias. The biostatistician is blinded to treatment modality to avoid bias in data analysis, with data labeled as "treatment modality 1" and "treatment modality 2" in the Excel sheet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Split-Mouth Design (Experimental): Our study involves comparing two different dental treatment modalities, the SMART Hall technique and standard Stainless Steel Crown (SSC) restoration, in a split-mouth design. In this design, each participant serves as their own control, receiving both interventions sequentially. The 'Single Arm' model aligns with our study structure, indicating that all participants receive both treatment modalities. This approach is consistent with our split-mouth study design, where each participant acts as their own control.
  Interventions: Procedure: SMART Hall Technique or procedure

INTERVENTIONS:
Procedure: SMART Hall Technique or procedure — The SMART Hall technique, a minimally invasive approach in pediatric dentistry for managing caries in primary teeth, involves gentle cavity preparation using hand instruments and minimal local anesthesia. A glass ionomer cement is used for restoration, followed by crown adaptation and cementation. Postoperative care and follow-up assessments at 3 and 6 months are included.
  The Stainless Steel Crown (SSC) technique for restoring extensively decayed primary molars involves tooth preparation, crown selection, adaptation, and cementation. Postoperative care and follow-up assessments at 3 and 6 months are also part of the procedure.
  Other Names: Conventional Stainless Steel Crown restoration

SUMMARY:
Dental caries, particularly in primary molars, significantly affects children's oral health and overall well-being. Traditional management with stainless steel crowns (SSCs) involves significant tooth reduction and advanced dental skills. Introduced in the 1970s, the Hall technique offers a less invasive alternative, minimizing tooth reduction compared to SSCs.

The SMART Hall technique represents a further evolution, emphasizing atraumatic cavity preparation using hand instruments. It offers advantages like minimal or no tooth reduction, minimized discomfort, improved patient cooperation, shorter treatment times, and cost-effectiveness.

Silver Diamine Fluoride (SDF) emerges as a promising non-invasive approach for managing dental caries in primary teeth, though it may cause temporary tooth discoloration. However, comparative evaluation with traditional SSC restorations remains limited.

To address this gap, a randomized clinical trial will evaluate the treatment outcomes of the SMART Hall technique versus conventional SSC restoration for managing occluso-proximal carious lesions (ICDAS CODE 3/4/5) in primary molars of young patients. Children aged 3 to 9 years requiring restorations will be included, assessing clinical outcomes, treatment time duration, and radiographical outcomes of both techniques at specific follow-up intervals of 3 months & 6 months.

This split mouth study will explore Clinical outcomes, radiographical outcomes, treatment time duration, and patient's pain perception with the chosen treatment modality. The findings will provide insights into the effectiveness and feasibility of the SMART Hall technique compared to the traditional SSC approach, informing evidence-based decision-making in pediatric dentistry and influencing treatment recommendations for preserving the health and function of primary molars in young children.

DETAILED DESCRIPTION:
AIM OF THE STUDY The aim of this research study is to compare the treatment outcomes of the SMART Hall technique with conventional stainless steel crown (SSC) restoration for managing occluso-proximal carious lesions (ICDAS CODE 3/4/5) in primary molars of 3- to 9-year-old children.

OBJECTIVES OF THE STUDY

1. To evaluate and compare the clinical success rates of the SMART Hall technique and conventional SSC restoration in managing occluso-proximal carious lesions in primary molars over a follow-up period of 3 & 6 months.
2. To evaluate and compare the treatment time duration of the SMART Hall technique and conventional SSC restoration in managing occluso-proximal carious lesions in primary molars.
3. To assess and compare the survival rates of teeth restored using the SMART Hall technique and conventional SSC restoration over a follow-up period of 3 & 6 months.
4. To assess and compare the radiographical outcomes of teeth restored using the SMART Hall technique and conventional SSC restoration over a follow-up period of 3 & 6 months.
5. To analyze and compare patient-reported perceptions of treatment using a Visual Analogue Scale between the two treatment modalities.

INCLUSION CRITERIA

1. Children aged 3 to 9 years old.
2. Presence of occluso-proximal carious lesions (ICDAS CODE 3/4/5) in one or more primary molars, confirmed through clinical examination and radiographic assessment.
3. Requirement for restorative treatment in the form of either the SMART Hall technique or conventional stainless steel crown (SSC) restoration, as determined by clinical assessment.
4. Willingness and ability of the parent/guardian to provide informed consent and ensure the child's attendance at follow-up appointments.
5. Adequate cooperation of the child during dental treatment and evaluation procedures, as determined by the clinician.

EXCLUSION CRITERIA

1. Presence of severe systemic medical conditions (e.g., uncontrolled diabetes, immunodeficiency disorders) that may compromise treatment outcomes or pose risks during dental procedures.
2. Use of medications known to interfere with dental treatment or healing, such as anticoagulants or immunosuppressants, unless medically managed and deemed safe by the treating healthcare provider.
3. History of adverse reactions to dental materials or procedures that may contraindicate participation in the study.
4. Inability of the child to tolerate local anesthesia or undergo dental treatment due to psychological, behavioral, or developmental factors.
5. Presence of extensive dental caries or additional oral pathologies requiring urgent or specialized dental care beyond the scope of the study.

METHODOLOGY Patients attending the Department Pedodontics & Preventive Dentistry department will be screened for identifying patients who fit into the inclusion & exclusion criteria. A total of 50 patients will be listed accordingly. Patients' parents / Guardian will be explained about the research study and treatments involved. Further, 25 patients will be randomly selected according to the determined sample size. Additional 5 patients will be recruited keeping in my the possibility of case attrition. A simple random selection method will be employed using Microsoft Excel program to generate patient pool to participate in this split mouth study.

Sampling method:

Probability sampling method, Simple Random sampling method using random number generators (RNGs)

Blinding:

Patients, Biostatistician and trained clinicians involved in evaluating clinical and radiographical outcomes will be kept blind about the type of treatment done in which primary tooth.

Training of examining clinicians:

To standardize the methods for training examiners in assessing clinical and radiographical outcomes, following steps will be followed:

1. Standardized protocol: These will outline the criteria and methods for assessing clinical and radiographical outcomes.
2. Training sessions: Conducting training sessions for the examiners to familiarize them with the standardized protocols.
3. Practice cases: Providing examiners with practice cases to assess using the standardized protocol.
4. Calibration exercises: Conducting calibration exercises to assess inter-examiner and intra-examiner variability. In these exercises, multiple examiners independently assess the same set of cases using the standardized protocol.

Assessing inter-examiner and intra-examiner variability: Intraclass Correlation Coefficient (ICC) statistical test will be employed to check for both inter-examiner and intra-examiner variability.

Blinding of biostatistician: Blinding the biostatistician to the type of treatment modality to minimize potential bias in data analysis. Providing data labeled as "treatment modality 1" and "treatment modality 2" in the Excel sheet effectively conceals the treatment assignment from the biostatistician.

Criteria for Clinical Assessment are as follows:

Successful

* Restoration appears satisfactory. No intervention required.
* No clinical sign or symptom of pulpal pathology
* No pulpal pathology visible on X-Ray.
* Tooth exfoliated

Minor failure

* Crown loss and tooth restorable
* Crown perforation
* Marginal caries
* Reversible pulpitis.

Major failure

* Irreversible pulpitis
* Dental abscess
* Crown loss and tooth is unrestorable
* Periradicular radiolucency

Clinical Parameters used in assessment are as follows:

* Pain - Present / Absent
* Mobility - Present / Absent
* Tender on percussion - Present / Absent
* Abscess or Sinus - Present / Absent

Radiographical Parameters used in assessment are as follows:

* No abnormal findings - Present / Absent
* Root resorption - Present / Absent
* Periapical pathology - Present / Absent
* Internal resorption - Present / Absent
* Furcation involvement - Present / Absent

The Visual Analogue Scale (VAS) will be utilized to evaluate patients' treatment experience.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 3 to 9 years old.
2. Presence of occluso-proximal carious lesions (ICDAS CODE 3/4/5) in one or more primary molars, confirmed through clinical examination and radiographic assessment.
3. Requirement for restorative treatment in the form of either the SMART Hall technique or standard stainless steel crown (SSC) restoration, as determined by clinical assessment.
4. Willingness and ability of the parent/guardian to provide informed consent and ensure the child's attendance at follow-up appointments.
5. Adequate cooperation of the child during dental treatment and evaluation procedures, as determined by the clinician.

Exclusion Criteria:

1. Presence of severe systemic medical conditions (e.g., uncontrolled diabetes, immunodeficiency disorders) that may compromise treatment outcomes or pose risks during dental procedures.
2. Use of medications known to interfere with dental treatment or healing, such as anticoagulants or immunosuppressants, unless medically managed and deemed safe by the treating healthcare provider.
3. History of adverse reactions to dental materials or procedures that may contraindicate participation in the study.
4. Inability of the child to tolerate local anesthesia or undergo dental treatment due to psychological, behavioral, or developmental factors.
5. Presence of extensive dental caries or additional oral pathologies requiring urgent or specialized dental care beyond the scope of the study.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Successful | Clinical success and survival rates of the procedure will be assessed at specific follow-up intervals of 3 months & 6 months.
  1. Restoration Satisfactory: The restoration appears satisfactory upon clinical examination, with no visible defects or issues.
     - No Intervention Required: The tooth does not require any additional intervention post-restoration.
  2. Absence of Pulpal Pathology:
     * No Clinical Signs or Symptoms of Pulpal Pathology: The patient exhibits no clinical signs or symptoms indicative of pulpal pathology, such as pain, swelling, or sensitivity.
     * No Pulpal Pathology Visible on X-Ray: Radiographic evaluation shows no signs of pulpal pathology, such as radiolucency or periapical lesions.
  3. Tooth Exfoliation:
     * Natural Tooth Exfoliation: The tooth exfoliates naturally, without the need for extraction.

SECONDARY OUTCOMES:
Minor failure | Clinical success and survival rates of the procedure will be assessed at specific follow-up intervals of 3 months & 6 months.
  1. Crown Loss and Tooth Restorable:
     * Measurement Tool: Clinical examination
     * Description: Assessment of the presence or absence of crown loss where the tooth remains restorable.
  2. Crown Perforation:
     * Measurement Tool: Clinical examination and radiographic evaluation
     * Description: Assessment of the integrity of the crown, specifically checking for any perforations.
  3. Marginal Caries:
     * Measurement Tool: Clinical examination and radiographic evaluation
     * Description: Detection of caries at the margins of the crown.
  4. Reversible Pulpitis:
     * Measurement Tool: Clinical examination, patient symptom reporting, and possibly radiographic evaluation
     * Description: Diagnosis of reversible pulpitis based on clinical signs and symptoms, such as pain that is not spontaneous and is relieved by analgesics or other treatment.
Major failure | Clinical success and survival rates of the procedure will be assessed at specific follow-up intervals of 3 months & 6 months.
  1. Irreversible Pulpitis:
     * Measurement Tool: Clinical examination, patient symptom reporting, and radiographic evaluation
     * Description: Diagnosis of irreversible pulpitis, characterized by persistent spontaneous pain not relieved by analgesics, confirmed through clinical and radiographic assessments.
  2. Dental Abscess:
     * Measurement Tool: Clinical examination and radiographic evaluation
     * Description: Identification of a dental abscess, indicated by swelling, pus discharge, and radiographic evidence of infection.
  3. Crown Loss and Tooth Unrestorable:
     * Measurement Tool: Clinical examination
     * Description: Assessment of crown loss where the tooth is deemed unrestorable, confirmed through clinical examination.
  4. Periradicular Radiolucency:
     * Measurement Tool: Radiographic evaluation
     * Description: Detection of periradicular radiolucency, indicating potential periapical pathology, as observed in radiographic images.

CONTACTS AND LOCATIONS:
Overall Officials: Saraswathi Bai Pakkirawadi Katika, M.D.S, Principal Investigator — Post Graduate Student in Department of Pediatric Dentistry & Preventive Dentistry
Locations (1):
- Dr Pakkirawadi Katika Saraswathi Bai, Tirupati, Andhrapradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Relevant masked IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from November 2025 until March 2026.
Access Criteria: Access on request to only researchers.
URL: https://vivli.org/

REFERENCES:
- [Background] Ayedun OS, Oredugba FA, Sote EO. Comparison of the Treatment Assessments of the Conventional Stainless-Steel Crown Restorations and the Hall Technique. West Afr J Med. 2020 Jul-Aug;37(3):253-259. PMID 32476119
- [Background] Ayedun OS, Oredugba FA, Sote EO. Comparison of the treatment outcomes of the conventional stainless steel crown restorations and the hall technique in the treatment of carious primary molars. Niger J Clin Pract. 2021 Apr;24(4):584-594. doi: 10.4103/njcp.njcp_460_20. PMID 33851682
- [Background] Ludwig KH, Fontana M, Vinson LA, Platt JA, Dean JA. The success of stainless steel crowns placed with the Hall technique: a retrospective study. J Am Dent Assoc. 2014 Dec;145(12):1248-53. doi: 10.14219/jada.2014.89. PMID 25429038